CLINICAL TRIAL: NCT06654479
Title: The Effect of Location and Duration of Nursing Interventions on Body Temperatures of Infants in the Neonatal Intensive Care Unit
Brief Title: The Effect of Nursing Interventions on Body Temperatures of Infants
Status: Completed | Type: Observational
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Beste Ozguven Oztornaci, Assist. Prof. Dr., Izmir Katip Celebi University
Other Study IDs: 22.09.2022/0380
Record Dates: First submitted 2024-10-20; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Hypothermia, Newborn
Keywords: Nursing; Newborn; Hypothermia
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The study included neonates treated in the neonatal intensive care unit.: In the newborns in the study, changes in body temperatures during routine nursing interventions of the nurses of the clinic were examined.
  Interventions: Other: In the newborns in the study, changes in body temperatures during routine nursing interventions of the nurses of the clinic were examined.

INTERVENTIONS:
Other: In the newborns in the study, changes in body temperatures during routine nursing interventions of the nurses of the clinic were examined. — The study is an observational study. The newborns were not intervened by the researcher. Body temperature changes were observed during routine practices of nurses in the clinic.

SUMMARY:
Aim: This study planned the intervention and care of term and preterm newborns treated in neonatal intensive care units, including thermoregulation, procedure duration and care with the opening technique of incubator covers.

Method: This non-participatory observational study was conducted between October 2022 and December 2023 with a total of 104 term and preterm newborns who were being treated in the Neonatal Intensive Care Unit of S.B.U. Dr. Behçet Uz Children's Diseases and Surgery Training and Research Hospital, Izmir, Turkey. In the study, the Case Report Form prepared by the researcher and based on the research method, dependent/independent variables and inclusion/exclusion criteria was used to collect data. The opening techniques of incubator lids were determined as double intervention window open, single intervention window open and incubator lid fully open. After selected newborns who met the inclusion/exclusion criteria, standardisation was ensured by explaining to the nurse who would provide care and intervention the location of the heat probe (right abdominal region) and that the patient should be in the supine position. The incubator temperature, incubator humidity, body temperature and neonatal intensive care room temperature and humidity before the procedure, the technique of opening the incubator lid during the care delivery phase and the intervention applied were recorded on the Case Report Form.

DETAILED DESCRIPTION:
Aim: This study planned the intervention and care of term and preterm newborns treated in neonatal intensive care units, including thermoregulation, procedure duration and care with the opening technique of incubator covers.

Method: This non-participatory observational study was conducted between October 2022 and December 2023 with a total of 104 term and preterm newborns who were being treated in the Neonatal Intensive Care Unit of S.B.U. Dr. Behçet Uz Children's Diseases and Surgery Training and Research Hospital, Izmir, Turkey. In the study, the Case Report Form prepared by the researcher and based on the research method, dependent/independent variables and inclusion/exclusion criteria was used to collect data. The opening techniques of incubator lids were determined as double intervention window open, single intervention window open and incubator lid fully open. After selected newborns who met the inclusion/exclusion criteria, standardisation was ensured by explaining to the nurse who would provide care and intervention the location of the heat probe (right abdominal region) and that the patient should be in the supine position. The incubator temperature, incubator humidity, body temperature and neonatal intensive care room temperature and humidity before the procedure, the technique of opening the incubator lid during the care delivery phase and the intervention applied were recorded on the Case Report Form. The researcher monitored the duration of the procedure with a chronometer at the beginning of the procedure. Body temperature, incubator temperature.

ELIGIBILITY:
Inclusion Criteria:

* In the neonatal intensive care unit,
* History of mature and premature birth (≤37 GH),
* Definitive diagnosis known,
* Newborns treated in a single brand of incubator, as different brands of incubators may vary in opening the lids and heating the incubators according to the characteristics of the incubator.

Exclusion Criteria:

* Diagnosed with asphyxia and receiving therapeutic cooling treatment,
* Within 10 days postoperatively,
* Active fever or a diagnosis of sepsis,
* Intervened under the radiant heater,
* Clinical condition deteriorated during the study period,
* Newborns who are followed and clothed to be placed with their mother.

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 104 newborns cared for by 72 nurses who consented to participate in the study and who met the inclusion criteria were included in the sample. No case was lost at the end of the study. The power level of the sample was found to be 0.878.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-02-08 (Actual)

PRIMARY OUTCOMES:
Body temperature of newborns | The study was completed in 17 months.
  Changes in body temperature of neonates during routine interventions by nurses

CONTACTS AND LOCATIONS:
Locations (1):
- İzmir Katip Çelebi University, Izmir, Çi̇ğli̇, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided